CLINICAL TRIAL: NCT06397937
Title: The SDOH-Homecare Intervention Focus Team (SHIFT) Trial to Mitigate Social Determinants of Stroke Outcomes and Build Community Capacity (The SHIFT Trial)
Brief Title: SDOH-Homecare Intervention Focus Team (SHIFT) Trial to Improve Stroke Outcomes
Acronym: SHIFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Olajide Williams, Professor of Neurology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ACYY0520; U01NS135533 (NIH); AAAV1743 (Other: Columbia University Irving Medical Center Institutional Review Board)
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Stroke; Social Determinants of Health
Keywords: stroke; social determinants of health; health disparities; community health workers; home visits
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Phase 3, randomized, blinded outcome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The SHIFT intervention team, comprising a community health worker (CHW), community social worker (CSW), and community nurse (CN),will make a first home visit within 72 hours of hospital discharge, and make regular visits to address SDOH barriers identified for each patient, provide individualized counseling, and assist with medication management, risk factor control, and health literacy.
  Interventions: Behavioral: SHIFT team intervention
- Usual Care (No Intervention): All patients will be given standard discharge information, including culturally/racially sensitive stroke education materials for post-stroke care, signs and symptoms of acute stroke, and management of stroke risk factors. Homecare referrals and other rehabilitation services will continue to be provided to discharged patients according to standard-of-care and treating physician referrals. Follow up clinic appointments at 4-6 weeks post discharge will be made with a stroke neurologist per clinical protocol. Thus the only difference between intervention and usual care will be the SHIFT intervention.

INTERVENTIONS:
Behavioral: SHIFT team intervention — The SHIFT team, comprising a community health worker (CHW), community social worker (CHW), and community nurse (CN) will visit the participant starting within 72 hours of hospital discharge and provide social service referrals related to food insecurity, housing, immigration, and employment, and assist with medical appointment preparation (CHW), deliver individualized counseling focused on coping skills, reducing caregiver strain, and the psychological distress associated with experiences of racism and SDOH (CSW), and address health literacy and review of treatment goals and medications (CN).
  Arms: Intervention

SUMMARY:
Primary Goal:

To test the hypothesis that among stroke patients 18-75 years with ≥3 SDOH risk factors, SHIFT will improve: (1) functional outcomes as measured by the SIS (Primary Outcome), (2) physiological outcomes as measured by changes in blood pressure and cognition, (secondary outcomes) and (3) epigenetic allostatic load biomarkers (exploratory outcome) such as DNA methylation (DNAm) and telomere length, at 6 months and 1-year post-stroke, compared with usual care (UC).

DETAILED DESCRIPTION:
Adverse Social Determinants of Health (SDOH) have been shown increase stroke risk in a dose dependent manner. The SDOH-Homecare Intervention Focus Team (SHIFT) trial is a Phase 3, randomized, blinded outcome trial that tests the hypothesis that a homecare intervention shortly after discharge from an acute stroke unit by a team comprising a community health worker (CHW), a community social worker (CSW) and a community nurse (CN) can improve health outcomes among stroke patients with three or more SDOH compared with UC.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke (arterial subtypes) or primary intracerebral hemorrhage (excluding diagnosis of probable cerebral amyloid angiopathy by Boston Criteria)
* African American/Black or Hispanic race-ethnicity
* Age 18-75 years old
* Have at least 3 SDOH barriers from within the 5 SDOH domains (Social and Community, Education, Economic, neighborhood/environment, Health Care)
* Have a discharge plan to 1) home with or without home services, or 2) acute rehabilitation with plan to return home after
* Pre-stroke Modified Rankin Scale score of ≤3
* Residence in New York City.
* English or Spanish speaking.
* Can provide informed consent and engage in the initial assessment prior to stroke discharge
* Lives in a household with a telephone, and has a caregiver (family member or Home Health Aide) if not fully independent on discharge. If the patient requires a family member to assist with activities of daily living or decision-making, the family member must state a willingness to be present at home visits where their assistance is needed.

Exclusion Criteria:

* Discharge disposition to a long-term care facility.
* Diagnosis of dementia or other neurological diagnosis that affects cognition
* Diagnosis of active major depression
* Aphasia severe enough to preclude initial examination
* Impaired level of consciousness at initial cognitive assessment
* Subarachnoid hemorrhage
* Diagnosis of probable cerebral amyloid angiopathy by Boston criteria
* Life expectancy less than 1 year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Stroke Impact Scale v3.0 | baseline, 6 months and 1 year
  a validated measure of disability and health-related quality of life after stroke

SECONDARY OUTCOMES:
Blood pressure | baseline, 6 months and 1 year
  change in blood pressure from baseline
cognition | baseline, 6 months and 1 year
  Montreal Cognitive Assessment battery (MoCA)
Stroke Specific Quality of Life (SSQOL) | 6 months and 1 year
  validated quality of life measure

OTHER OUTCOMES:
Medication Adherence | 6 months and 1 year
  medication adherence
30-day readmission rate | 30 days post discharge
  incidence of readmission to the hospital within 30 days of discharge
Epigenetic biomarkers of stress | baseline, 6 months and 1 year
  DNA methylation, telomere length

CONTACTS AND LOCATIONS:
Overall Officials: Olajide Williams, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
To share individual participant data (IPD) of baseline characteristics, follow up, outcomes, etc. based on NIH/NINDS requirements.
Supporting Information: Study Protocol
Time Frame: As per NIH/NINDS requirements
Access Criteria: All items required by NIH/NINDS will be publicly shared.

REFERENCES:
- [Background] Harris J, Boehme A, Chan L, Moats H, Dugue R, Izeogu C, Pavol MA, Naqvi IA, Williams O, Marshall RS. Allostatic load predicts racial disparities in intracerebral hemorrhage cognitive outcomes. Sci Rep. 2022 Oct 3;12(1):16556. doi: 10.1038/s41598-022-20987-x. PMID 36192526
- [Background] Mallaiah J, Williams O, Allegrante JP. Development and Validation of a Stroke Literacy Assessment Test for Community Health Workers. Health Educ Behav. 2024 Oct;51(5):764-774. doi: 10.1177/10901981241245050. Epub 2024 Apr 22. PMID 38646736